CLINICAL TRIAL: NCT06224322
Title: Evaluation of Factors Affecting Caregiver Burden in Cerebral Palsy Patients Undergoing Hip and Knee Surgery
Brief Title: Caregiver Burden in Cerebral Palsy Undergoing Hip and Knee Surgery
Acronym: Caregiver CP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, AHMET MUCTEBA YILDIRIM, Principal Investigator, Istanbul University
Other Study IDs: 2234234
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy; Care Giving Burden
MeSH Terms: conditions — Cerebral Palsy; Caregiver Burden | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cerebral Palsy Patients Parent: Parents of patients who underwent knee and hip surgery for cerebral palsy
  Interventions: Other: Assesment Scale

INTERVENTIONS:
Other: Assesment Scale — Caregiving burden will be assessed with Turkish validated scoring tools such as the Zarit scale and the Pediatric Quality of Life Inventory (PEDSQL) Family Impacts module before and after surgery.
  Other Names: Questionnaire

SUMMARY:
The aim of this observational study was to obtain information about the change in the burden of care of parents of children with cerebral palsy after hip and knee surgeries. The main questions it aims to answer are:

Q1-Does caregiver burden change after hip and knee surgeries? Q2-If so, which factors contribute more positively to this situation? Participants will be asked to answer the scales given to them periodically before and after the surgery.

DETAILED DESCRIPTION:
One of the most common causes of disability in childhood is cerebral palsy, which develops due to damage to the central nervous system. Children diagnosed with cerebral palsy face different problems in every period of their lives. The child, his/her family and the society he/she lives in should be considered as a whole. There is a mechanism that mutually affects each other.

Parenting, caring for and living with a child with cerebral palsy can have many negative effects on the lives of parents and create additional burdens for them. Parents may have to choose between their own needs, the needs of other members of the family and the needs of the child with cerebral palsy, and may spend most of their time with their disabled child. This can negatively affect the burden, stress level, physical activity level, quality of life, psychological status and self-efficacy perception.

The primary aim of this study is to evaluate the caregiver burden in Cerebral Palsy, which is the most common cause of morbidity in the pediatric age group in orthopedics, and to analyze the factors that negatively affect it. Our hypothesis is that the functional mobilization status of patients will increase, especially as a result of hip surgeries, reducing caregiver burden.

ELIGIBILITY:
Inclusion Criteria:

1. Parent Age

   a. Being in the 20-60 age group.
2. Diagnosis

   1. Having a child with clinically diagnosed cerebral palsy
   2. The movement scale of the cerebral palsy patient is between GMFS 3 and 5
3. A minimum follow-up of 12 months after surgery
4. The primary carer is the mother or father

Exclusion Criteria:

1. The patient and his/her family have been lost to follow-up
2. Having another disabled person in need of care in the family
3. Family's unwillingness to participate in the study
4. Loss of a parent

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Our study will be conducted with the parents of children with cerebral palsy who are admitted to the Orthopaedics Unit of Istanbul Medical Faculty and will be operated on in the knee-hip region.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Zarit Caregiven Burden scale | Preoperative, Postoperative three, six and twelve month
  The 22-item instrument is included in this scale. Each item in the questionnaire is a statement that the carer is asked to confirm using a 5-point scale. The answer options range from 0 (Never) to 4 (Almost Always).

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory (PEDSQL) Family Impacts module | Preoperative, Postoperative three, six and twelve month
  This scale was developed by James James in 2004 to measure the effects of a child with an illness on family functioning. It was developed by Varni. It consists of 6 sub-factors and 36 statements. Physical Functioning (6 items), 2) Emotional Functioning (5 items), 3) Social Functioning (4 items), 4) Cognitive Functioning (5 items), 5) Communication (3 items), 6) Concern (5 items) and 2 subscales measuring parent-reported family functioning; 7) Daily Activities (3 items) and Family Relationships (5 items).

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet MD Demirel, MD, Principal Investigator — Assistant Professor
Locations (2):
- Turkey (Türkiye) (2):
  - Department of Orthopaedics and Traumatology, Istanbul University, Istanbul, Turkey, Istanbul, Fatih-Topkapı
  - Istanbul Unıversity Medicine Faculty Orthopaedic Department, Istanbul, Fatih

IPD SHARING:
Plan to Share IPD: No
Maybe one year later ı am going to share ıpd